CLINICAL TRIAL: NCT07371377
Title: The TOF3D Mechanomyograph. Evaluation of a New Device for Assessment of the Neuromuscular Block.
Acronym: MMG versus AMG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Hersfeld-Rotenburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MMG and TOF3D
Record Dates: First submitted 2026-01-10; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Mechanomyography; Neuromuscular Blockade Monitoring
Keywords: mechanomyography; tetanic fade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- comparison of mechanomyograph and acceleromyograph (Other)
  Interventions: Device: measurement of the time course of a neuromuscular block
- comparison of tetanic fade versus train of four ratio (Other)
  Interventions: Device: measurement of the time course of a neuromuscular block

INTERVENTIONS:
Device: measurement of the time course of a neuromuscular block — a new device is compared to an established one.

SUMMARY:
In clinical anesthesiologic practice, most institutions use acceleromyography in order to assess the degree of a neuromuscular block.

The aim of the present study is to assess a new device using mechanomyography. Until recently, this method was reserved for experimental settings. It seems to be able to work more precisely, and additionally, it offers the opportunity to use other stimulation patterns than acceleromyographic measurements.

The investigation is divided into two parts:

Part 1 compares the mechanomyograph directly with an acceleromyograph. In part 2, two mechanomyographs using different stimulation patterns are compared with each other.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for surgery requiring general anesthesia with neuromuscular blocking agents

Exclusion Criteria:

* anticipated or known difficult airway
* increased risk for aspiration
* pregnancy
* neuromuscular disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
difference in time to recovery to a train of four ratio of 1,0. | from enrollment to the end of anesthesiologic treatment at the day of surgery (2-3 weeks after enrollment)
  difference in time to recovery to a train of four ratio of 1,0 measured by acceleromyography and mechanomyography, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and Intensive Care Medicine, Bad Hersfeld, Germany

IPD SHARING:
Plan to Share IPD: No